CLINICAL TRIAL: NCT01717495
Title: Thromboembolic Complications Associated With Pacemaker or Implantable Cardioverter-Defibrillator Procedures: a Prospective Registry
Brief Title: Thromboembolic Complications After Pacemaker or Implantable Cardioverter-Defibrillator Procedures
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Duke University (Other)
Responsible Party: Principal Investigator, Roberto Costa, Associated Professor of Cardiovascular Surgery, MD PhD, University of Sao Paulo
Other Study IDs: CAPPesq: 0730/11
Record Dates: First submitted 2012-09-30; First posted 2012-10-30 (Estimated); Last update posted 2013-05-07 (Estimated); Status verified 2013-05

CONDITIONS: Bradyarrhythmias; Arrhythmias; Cardiovascular Disease; Venous Thrombosis; Pulmonary Embolism
Keywords: Pacemaker; Implantable-cardioverter defibrillator; Cardiac Pacing, Artificial/adverse effects; Venous thrombosis; Pulmonary embolism; Phlebography; Biological markers; Computed tomography angiography
MeSH Terms: conditions — Bradycardia; Arrhythmias, Cardiac; Cardiovascular Diseases; Venous Thrombosis; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood Fibrinogen, D Dimer, Antithrombin, Prothrombin fragment 1 +2, thromboxane B, Platelets, Plasminogen
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Implantation Procedures: Patients submitted to initial pacemaker or ICD implantation
- Reoperation Procedures: Patients submitted to pacemaker or implantable cardioverter-defibrillator generator replacements, upgrade procedures and lead extraction

SUMMARY:
This is a large prospective registry of patients submitted to cardiac electronic devices implantation designed to investigate the incidence, risk factors and prognostic of thromboembolic complications associated with transvenous lead implantation.

DETAILED DESCRIPTION:
More than 235.500 cardiac pacemakers and cardioverter-defibrillators are implanted in the US every year, with an estimated 25,000 new implants in Brazil. Despite its proven clinical effectiveness and efficacy for a number of clinical conditions such as arrhythmias, the number of adverse events in the post-implant period remains substantial. Among these complications, venous obstructions occurs anywhere between 14% and 64% of all patients, causing devastating consequences such as upper extremity deep venous thrombosis and pulmonary embolism, ultimately leading to either significant impairment or death. Although retrospective studies have demonstrated the high incidence of these complications, as a consequence of a paucity of reliable registries we know next to nothing regarding how these venous lesions may influence the clinical outcome and mortality of patients, whether laboratorial markers may contribute to the early diagnosis of venous thrombosis and its complications, and about properties of diagnostic imaging for the identification of thromboembolic complications after permanent transvenous leads implantation.

The objective of this study is therefore to propose a significant improvement in an existing clinical database located within the Heart Institute (INCOR) at the University of Sao Paulo to enable the provision of answers to a clinical, biomarker, and imaging-related research questions. Specifically, our aims are to:

* Aim 1 - Registry infrastructure: In collaboration with professors from Duke University, we will create a series of improvements to the current database to enable it to serve as a platform not only for the current studies but also for future longitudinal, randomized studies. These include the standardization of variables in accordance with international guidelines, increase in patient retention and the ability to have additional data points in-between clinical appointments, improvement in the determination of cause of mortality, data quality monitoring, the creation of an item bank to measure aspects of quality of life that are specific for this population, as well as the integration of images and biomarkers to the clinical database.
* Aim 2 - Diagnostic imaging methods: To identify the incidence of upper extremity deep venous thrombosis after cardiac devices implantations or reoperation procedures, as well, the incidence of symptomatic and asymptomatic pulmonary thromboembolism.
* Aim 3 - Prognostic clinical factors: To study the impact of thromboembolic complications in the clinical prognostic and mortality of patients;
* Aim 4 - Prognostic biomarkers: To determine the association between the biomarkers related with alterations in the hemostasis system and the occurrence of venous thrombosis (biomarkers: Fibrinogen, D Dimer, Antithrombin, Prothrombin fragment 1 +2, thromboxane B, Platelets, Plasminogen)

At the end of this study we will have a registry with one of the largest number of patients with this condition around the world, fully equipped for future randomized controlled trials. We will also have a much better understanding regarding clinical, imaging, and biomarkers for this condition.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Pacemaker/ implantable-cardioverter defibrillator (ICD) / cardiac resynchronization therapy (CRT) initial implant by transvenous approach or
* Patients submitted to reoperation procedures, as: pulse generator replacement, implant of an additional lead, lead extraction, lead repositioning;
* Subject agreed to participate and signed the consent form

Exclusion Criteria:

* Patients with a history of venous thromboembolism, coagulopathy or malignancy
* Pregnancy
* Life expectancy of less than one year
* Contraindication to administration of iodinated contrast (creatinine > 3.0)
* Unable to attend the follow-up appointments

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Thromboembolic complications | Participants will be evaluated at 1, 6, 12 months after the surgical procedure
  Upper extremity deep venous thrombosis Pulmonary embolism All cause mortality

SECONDARY OUTCOMES:
Venous lesions | Participants will be evaluated at 12 months after the surgical procedure
  Venous stenosis (any degree) detected by subtraction venography

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Costa, MD PhD, Principal Investigator — University of Sao Paulo; Katia R Silva, RN PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Heart Institute (InCor) do Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo, Brazil